CLINICAL TRIAL: NCT03081819
Title: A Phase I Study of SH003 for Evaluate Safe Dose Range in Patients With Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Gyu Ko, Professor, Kyunghee University Medical Center
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ISEE_2015_SH003
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH003 (Experimental): Participant will take SH003 for 3 weeks.
  Interventions: Drug: SH003

INTERVENTIONS:
Drug: SH003 — Herbal medicine for cancer treatment

SUMMARY:
A Phase I study of SH003 for evaluate safe dose range in patients with solid cancer.

The first dose group receives SH003 for 3 weeks. If the adverse events occur in less than one in six participants, the dose is escalated.

The second dose group receives SH003 for 3 weeks. If the adverse events occur in less than one in six participants, the dose is escalated.

The third dose group receives SH003 for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Patients with histologically and cytologically confirmed solid tumor
* Patients who have failed standard treatments, such as previous chemotherapy or radiotherapy, or who are inoperable, refractory, or progressive.
* ECOG score 0-2
* Patients with a minimum life expectancy of 12 weeks at the scheduled starting date of the study drug
* Previous treatment with surgery or radiotherapy, at least 4 weeks since end of treatment is allowed (the patient should have been recovered from any side effects.
* Patients who can swallow pills.
* Patients who provide written informed consent for participation in the trial

Exclusion Criteria:

* Known hypersensitivity to any study drug component, including Astragalus membranaceus, Angelica gigas, or Trichosanthes Kirilowii Maximowicz
* Patients with pre-existing cardiac conditions:
* Prior documented myocardial infarction within the last 6 months
* Pre-existing cardiac failure (NYHA class III-IV)
* Atrial fibrillation on anti-coagulants
* Unstable angina
* Severe valvulopathy
* Cardiac angioplasty or stenting with in the last 6 months
* Pregnant or lactating females
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety
* Active uncontrolled infection, including known history of AIDS or hepatitis B or C
* Any psychological, sociological, or geographical condition that could potentially interfere with compliance with the study protocol
* Concurrently receiving any other investigational agents while on study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3 weeks
  Grade 3-4 adverse event using CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheon C, Ko SG. A Phase I Study to Evaluate the Safety of the Herbal Medicine SH003 in Patients With Solid Cancer. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420911442. doi: 10.1177/1534735420911442. PMID 32186413
- [Derived] Cheon C, Kang S, Ko Y, Kim M, Jang BH, Shin YC, Ko SG. Single-arm, open-label, dose-escalation phase I study to evaluate the safety of a herbal medicine SH003 in patients with solid cancer: a study protocol. BMJ Open. 2018 Aug 5;8(8):e019502. doi: 10.1136/bmjopen-2017-019502. PMID 30082340